CLINICAL TRIAL: NCT03961763
Title: Effect of n-3 Fatty Acid Supplementation in Hyperlipidemic Patients Taking Statins, on Lipid Profile, Including Small Dense LDL: A Randomized, Placebo-controlled, Double-blind Trial.
Brief Title: Effect of n-3 Fatty Acid Supplementation in Hyperlipidemic Patients Taking Statins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1288/17/GD/CSN
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Cardiovascular Diseases; Hyperlipidemias; Dyslipidemias
Keywords: omega-3; EPA; DHA; sdLDL; cardiovascular disease; hyperlipidemia; dyslipidemia
MeSH Terms: conditions — Cardiovascular Diseases; Hyperlipidemias; Dyslipidemias | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- omega-3 supplement (Active Comparator): This group will receive a daily dose of 4g EPA+DHA (which is the recommended safe tolerable upper intake level of omega-3 supplements for healthy individuals) for eight weeks.
  Interventions: Dietary Supplement: EPA+DHA
- Placebo (Placebo Comparator): This group will receive a daily dose of 4g olive oil placebo for eight weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: EPA+DHA — 4 g/day EPA+DHA in tablets of 1g, 4 tablets daily, over 8 weeks (56 days)
  Other Names: marine omega-3; fish oil
  Arms: omega-3 supplement
Other: Placebo — 4 g/day olive oil placebo in tablets of 1g, 4 tablets daily, over 8 weeks (56 days).
  Other Names: Non-active ingredient
  Arms: Placebo

SUMMARY:
Epidemiological and clinical evidence suggests that high-dose intake of long-chain n-3 fatty acids have a favorable role in altering blood TG and non-HDL cholesterol when combined with statins in hyperlipidemic patients. Their efficacy in altering low density lipoprotein cholesterol particle size and concentration is yet to be confirmed.

This study evaluates the effects of adding 4/day eicosapentaenoic acid (EPA) + docosahexaenoic acid (DHA) to stable statin therapy on blood TG, non-HDL, LDL-C as well as small dense (sdLDL) particle concentration in a group of hyperlipidemic patients.

In this randomized, placebo-controlled, double-blind parallel group study, 44 subjects who were already on statin therapy for > 8 weeks and had non-HDL-C levels above the National Lipid Association Recommendations were randomized into two groups. For 8 weeks, together with their prescribed atorvastatin, the intervention group received 4g/day EPA+DHA (in ethyl ester form) while the control group received 4g/day olive oil (placebo). Baseline measurements of non-HDL-C, TG, TC, HDL-C, LDL-C, VLDL-C and sdLDL were repeated at week 8. Differences in dietary intake were assessed with a weighed 3-day food diary at week 4. Primary outcome measures are the percent change in non-HDL-C and sdLDL particle concentration from baseline to the end.

DETAILED DESCRIPTION:
This study is a parallel randomised, double-blind placebo - controlled trial which was conducted in Istanbul, Turkey.

BACKGROUND

Cardiovascular disease (CVD) has been, and still is the number 1 cause of deaths all over the world. According to the World Health Organisation (WHO), 1 of every 3 death was caused by CVD in 2012. Heart disease and stroke were the No. 1 and No. 2 killers worldwide, according to American Heart Association. In Turkey, it is even worse, 40% of all deaths were caused by CVD. Such high prevalence naturally brings a huge disease burden and in many countries there are ongoing research to mitigate CVD risk.

It is essential to highlight that CVD is not a single disease, it is actually a family of diseases that mostly cause by a common pathology named "atherosclerosis". Atherosclerosis is plaque formation in artery walls which leads a reduced lumen diameter, causing organ damage or clinical events like myocardial infarction (MI), angina or stroke. One of the two reasons of atherosclerosis is hyperlipidemia, which is the theme of this study. Atherosclerosis and lipids are evident to be related; the elevations in circulating LDL cholesterol level plays a central role in atherogenesis, given the fact that they cause the formation of fatty plaque. Therefore, in all clinical guidelines, LDL level is the primary target to prevent atherosclerosis.However, more recent studies have revealed that LDL is structurally heterogeneous based on its size and density. There are large, buoyant LDL particles and small, dense LDL particles, which are believed to be more atherogenic. Individuals that have a large amount of small and dense LDL particles are at an increased risk of CV events, regardless of their total LDL level. In studies, small and dense LDL profile was associated with a three-fold to seven-fold increase in risk of CVD as they:1- Have the increased ability to penetrate arterial wall. 2- Are readily oxidized.

The main therapeutic approach to treat small&dense LDL is using drugs that lower serum triglyceride (TG) levels, as they also cause a change in the LDL size profile to larger, less dense and, therefore, less atherogenic species. Most commonly used such drugs are statins. Apart from statins, there is strong evidence that omega-3 fatty acids also have a beneficial effect in lowering TGs. However, their effect on small, dense LDL has not been studied enough yet. If omega-3 fatty acids have a beneficial effect in changing LDL profile to less dense and larger particles, omega-3 supplementation will be quite effective for patients with hyperlipidemia. Given the fact that statin use is the gold standard in all clinical guidelines, this study will not compare statins with omega-3 fatty acids and instead, compare statin monotherapy to the combined use of statin and omega-3 supplements to investigate whether omega-3 fatty acids have a supportive role to statin.

RECRUITMENT AND SAMPLING:

Eligible participants were men or women from Istanbul, Turkey, aged between 50 and 79 years who had been receiving a stable dose of atorvastatin for the control of LDL-C levels at least for 8 weeks before initial screening.

One hundred patients were selected for initial screening and 44 matched the inclusion/exclusion criteria and were randomized to the intervention using www.randomization.com.

Participants were informed informally via telephone first, and then invited to the Clinic by a Patient Invitation Letter. A structured one-to-one information session was carried out with each participant at the Clinic, during which they were given a Participant Information Sheet. Participants provided written informed consent by signing the a Participant Consent Form.

SAMPLE-SIZE

Total sample size was 44, consisting of two 22-subject groups (control and intervention group).

A targeted sample size of 36 subjects (18 per arm) was expected to provide at least 80% power to detect a difference of 5% or above in primary outcome non-HDL-C and LDL-C III particle concentration when compared with placebo (α=0.05) . Sample size was assigned as 44 to allow for subject attrition and other potential causes of study withdrawal up to 20%.

The power calculation was based on the mean changes in non-HDL-C measurement of the previous COMBOS trial which is a largest randomized placebo controlled trial that has the same design with this study. Data from COMBOS trial is summarized as follows:

Intervention Group:

baseline non-HDL mean + standard deviation (SD): 135.8 mg/dL + 24.5 mg/dL final non-HDL mean + SD: 124.1 mg/dL + 24.7 mg/dL Percent change: -7.9%

Placebo Group:

baseline non-HDL mean +SD: 141.3 mg/dL + 29.3 mg/dL final non-HDL mean + SD: 138.8 mg/dL + 32.0 mg/dL Percent change: -1.5%

METHODS

A randomized, double-blind, placebo controlled, parallel groups study was carried out. Before entry into the intervention phase of the study, 8-weeks of dietary lead-in was carried out. Study participants received dietary counselling for the 8 weeks before the intervention, based on the heart-healthy diet structured in the United Kingdom (UK) National Institute of Health Care Excellence (NICE) guidelines (2014) and were instructed to maintain this diet throughout the study. Adherence to dietary advice was also measured by a 3-day weighed intake food diary at Week 4. Household measures were used to assess the food intake. Nutrient content of the diet was estimated using Nutritics software (Nutritics Ltd, Ireland) using UK: Scientific Advisory Committee on Nutrition (SACN) 2015 food composition tables.

After the dietary lead-in, baseline measurements of fasting blood Triglycerides (TG), Total Cholesterol (TC), High-density Lipoprotein cholesterol (HDL-C), Low-density Lipoprotein cholesterol (LDL-C), and LDL-C sub groups (LDL-C I, LDL-C II, LDL-C III, LDL-C IV, LDL-C V) were carried out for all subjects at 2 clinics separated by 1 week, and the means were used as baseline values. Non-High-density Lipoprotein cholesterol (non-HDL-C) was calculated by subtracting HDL-C from TC.

After baseline measurements, all participants were randomized in equal numbers to receive either 4g/day EPA (75%) & DHA (25%) ethyl esters or 4g/day olive oil (placebo) for 8 weeks in combination with the same dose of atorvastatin they had been prescribed. For all subjects, atorvastatin dosage was kept constant throughout the trial.

Both groups consumed four 1000mg capsules orally 4 times daily and compliance was measured by the number of capsules consumed relative to the number estimated to be consumed.

Baseline measurements were repeated at the end of week 8. Study participants and investigators remained blinded to all laboratory results until completion of analysis.

BIOCHEMICAL MEASUREMENTS

Laboratory analyses were performed by e-Lab Laboratories (Istanbul, Turkey) on the serum or plasma of 12 hours fasting blood samples. LDL-C, VLDL-C and HDL-C was measured with homogeneous enzymatic colorimetric assay of Roche Diagnostics (USA). TG and TC was measured with enzymatic colorimetric assay of Roche Diagnostics (USA). LDL-C subgroups were analyzed with electrophoresis by Lipoprint (Quantimetrix, USA).

STATISTICAL ANALYSIS

Statistical analyses was be performed with Statistical Package for the Social Sciences (SPSS) version 24 (IBM, USA).

Demographic and baseline analysis was performed for all study participants, while efficacy analysis was performed only on subjects that successfully completed the 8-week study protocol. The primary efficacy end points are non-HDL and LDL-C III particle concentration percentage change from baseline; secondary efficacy end points are changes in TG, TC, LDL-C, VLDL-C and HDL-C.

Normal distribution of the sample was checked with Shapiro-Wilk's test. Mixed model ANOVA test was carried out to compare changes in outcome parameters from baseline to end-of-treatment between the intervention and control groups.

Paired t-tests were performed to analyze the changes from baseline to Week 8 for each outcome parameter, and multiple Independent t-tests were performed to analyze significant differences between groups across time points. A P-value < 0.05 determined statistical significance.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female, aged between 50 and 80
2. Current combined hyperlipidemia: people whose LDL and non-HDL levels are above the National Lipid Association recommendations according to their risk groups. non-HDL is also considered given the fact most recent research states looking at both values is a better risk indicator than looking at LDL alone. (Appendix 12: National Lipid Association Treatment Guideline)
3. Currently on statin prescription.

Exclusion Criteria:

1. Current use of n-3 supplements
2. Recent history of certain heart, kidney, liver, or cancer:

   Patients that have had any type of heart surgery, Patients that are diagnosed with any type of cancer and/or have had any kind of cancer therapy, Patients that have had kidney failure, Patients that have had liver failure, in the past 6 months
3. Pregnant or lactating females

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
small &dense LDL I | 0 and 8 weeks
  LDL-C III particle concentration (mg/dL)
non-HDL-C | 0 and 8 weeks
  non-HDL cholesterol (mg/dL)

SECONDARY OUTCOMES:
TG | 0 and 8 weeks
  blood Triglycerides (mg/dL)
TC | 0 and 8 weeks
  total blood cholesterol (mg/dL)
HDL-C | 0 and 8 weeks
  blood high density lipoprotein cholesterol (mg/dL)
LDL-C | 0 and 8 weeks
  blood low density lipoprotein cholesterol (mg/dL)
VLDL-C | 0 and 8 weeks
  blood very low density lipoprotein cholesterol (mg/dL)
large&buoyant LDL-C I | 0 and 8 weeks
  LDL-C I particle concentration (mg/dL)
large&buoyant LDL-C II | 0 and 8 weeks
  LDL-C II particle concentration (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Sohail Mushtaq, PhD, Principal Investigator — University of Chester
Locations (1):
- Pax Clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dogay Us G, Mushtaq S. N-3 fatty acid supplementation mediates lipid profile, including small dense LDL, when combined with statins: a randomized double blind placebo controlled trial. Lipids Health Dis. 2022 Sep 1;21(1):84. doi: 10.1186/s12944-022-01686-y. PMID 36050695